CLINICAL TRIAL: NCT01181310
Title: A Five-Period, Placebo-Controlled, Crossover Study to Evaluate the Effect of Donepezil and MK-3134 on Reversal of Cognitive Impairment Associated With a Single-Dose of Scopolamine.
Brief Title: Placebo-Controlled Crossover Study to Evaluate Donepezil and MK-3134 for Reversal of Cognitive Impairment Associated With Scopolamine Administration (3134-005)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3134-005; 2007-001894-27 (EudraCT Number)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Dementia
Keywords: dementia, cognitive impairment, neurodegeneration, Alzheimer's, acetylcholine, AchE
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Nerve Degeneration; Pain | interventions — Scopolamine; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- A, B, D, E, C (Experimental): Participants received treatment A, B, D, E, C for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- B, C, E, A, D (Experimental): Participants received treatment B, C, E, A, D for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- C, D, A, B, E (Experimental): Participants received treatment C, D, A, B, E for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- D, E, B, C, A (Experimental): Participants received treatment D, E, B, C, A for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- E, A, C, D, B (Experimental): Participants received treatment E, A, C, D, B for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- A, C, B, E, D (Experimental): Participants received treatment A, C, B, E, D for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- B, D, C, A, E (Experimental): Participants received treatment B, D, C, A, E for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- C, E, D, B, A (Experimental): Participants received treatment C, E, D, B, A for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- D, A, E, C, B (Experimental): Participants received treatment D, A, E, C, B for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg
- E, B, A, D, C (Experimental): Participants received treatment E, B, A, D, C for Periods 1, 2, 3, 4, and 5, respectively.
  Interventions: Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine; Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg; Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg; Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg; Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg

INTERVENTIONS:
Drug: A: Placebo to match Donepezil and MK-3134 + Placebo to match Scopolamine — Single doses of placebo to match both donepezil and MK-3134 PO, plus a single dose of placebo to match scopolamine SQ.
Drug: B: Placebo to match Donepezil and MK-3134 + Scopolamine 0.5 mg — Single doses of placebo to match both donepezil and MK-3134 PO, plus a single dose of scopolamine 0.5 mg SQ.
Drug: C: MK-3134 25 mg + Scopolamine 0.5 mg — A single dose of MK-3134 PO 25 mg, plus a single dose of scopolamine SQ 0.5 mg.
Drug: D: Donepezil 10 mg + Scopolamine 0.5 mg — A single dose of donepezil 10 mg PO, plus a single dose of scopolamine 0.5 mg SQ.
  Other Names: Aricept (donepezil)
Drug: E: Combo: Donepezil 10 mg + MK-3134 25 mg + Scopolamine 0.5 mg — A combination of single doses of all active drugs: donepezil 10 mg and MK-3134 25 mg PO, plus scopolamine, SQ.
  Other Names: Aricept (donepezil)

SUMMARY:
The drug, scopolamine, can result in short-term impairments of cognitive function, attention, and memory that resemble those seen in aging and Alzheimer's disease. This study tested the capability of both individual and combined doses of MK-3134 and the current standard treatment: donepezil (Aricept), to reverse such impairments, following a single dose of scopolamine. Participants were evaluated after each of 5 different treatment periods (in a cross-over, double-dummy design): A: placebo to match both donepezil (oral [PO]) and MK-3134 (PO) followed by placebo scopolamine (subcutaneous [SQ]); B: placebo to match both donepezil (PO) and MK-3134 (PO), followed by scopolamine SQ; C: MK-3134 (PO) followed by scopolamine SQ; D: donepezil (PO) followed by scopolamine SQ; E: MK-3134 (PO) and donepezil (PO) followed by scopolamine SQ. The doses of MK3134, donepezil, and scopolamine were the same over all treatment arms in which the specified drug was administered. There were 8 total visits for each treatment period, including 5 Treatment Visits requiring 14-day intervals between visits for study-drug washout. Participants were assessed for cognitive function before and after each treatment period during the Treatment Visits.

ELIGIBILITY:
Participants were eligible for inclusion in the study who were:

* Male between 18 and 40 years of age.
* Non-smokers, in good health (as defined in protocol), and were willing to follow study-related procedures.

Participants were not eligible for inclusion in the study if they:

* Had a history of illness that, in the opinion of the study investigator or as specified in protocol, might confound the results of the study or posed an potential, additional risk to the participant if they were to participate in the study.
* Were taking any medication (prescription, nonprescription, vitamin supplements or herbal, illicit or legitimate) except for acetaminophen.
* Had a history of any significant head injury/trauma.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
CogState Early Phase Battery, Groton Maze Learning Test (GMLT) as measured by the number of errors on the GMLT over time (area under the GMLT-time curve) over hours 1-12. | 1, 2, 3, 4, 6, 8, and 12 hours relative to administration of SQ scopolamine or SQ placebo
  Participants learned a hidden pathway through a maze (10 x 10 grid of tiles on a computer touch screen) using step-by-step guess, with trial and error feedback after each step. Once the pathway was learned, participants repeated the same pathway four more times. The number of pathway errors was used to indicate the level of cognitive function.

REFERENCES:
- [Derived] Cho W, Maruff P, Connell J, Gargano C, Calder N, Doran S, Fox-Bosetti S, Hassan A, Renger J, Herman G, Lines C, Verma A. Additive effects of a cholinesterase inhibitor and a histamine inverse agonist on scopolamine deficits in humans. Psychopharmacology (Berl). 2011 Dec;218(3):513-24. doi: 10.1007/s00213-011-2344-y. Epub 2011 Jun 7. PMID 21644059